CLINICAL TRIAL: NCT04734626
Title: Magnetic Resonance Imaging (MRI) Muscle Phenotyping in Mitochondrial Disease
Brief Title: CrCest Study in Primary Mitochondrial Disease
Status: Enrolling by invitation | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-016520; 1R01AR083552-01A1 (NIH)
Record Dates: First submitted 2021-01-25; First posted 2021-02-02 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Mitochondrial Diseases
MeSH Terms: conditions — Mitochondrial Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mitochondrial Disease: Individuals with suspected (based on clinical presentation) or definite genetic mitochondrial disease
  Interventions: Diagnostic Test: Creatine Chemical Exchange Saturation Transfer (CrCEST) Imaging Sequence
- Healthy Controls/Volunteers: Individuals with no history of suspected (based on clinical presentation) or definite genetic mitochondrial disease
  Interventions: Diagnostic Test: Creatine Chemical Exchange Saturation Transfer (CrCEST) Imaging Sequence

INTERVENTIONS:
Diagnostic Test: Creatine Chemical Exchange Saturation Transfer (CrCEST) Imaging Sequence — CrCEST be used to assess creatine distribution and concentrations in muscle (lower extremity), both at rest and after recovery from a brief foot-pedal depression exercise

SUMMARY:
The purpose of this study is to perform a "muscle phenotyping" magnetic resonance imaging (MRI) assessment in patients receiving clinical care at the Children's Hospital of Philadelphia (CHOP) for mitochondrial disease that is either suspected (based on clinical presentation) or has a definite genetic diagnosis. The MRI assessment quantifies skeletal muscle oxidative phosphorylation (OXPHOS) capacity.

Investigators hope that this study will contribute to our current knowledge of mitochondrial diseases and this study will help create a new diagnostic tool for use in both clinical care and in clinical trials.

DETAILED DESCRIPTION:
This research study visit will occur on the same day as the participants clinically scheduled MRI. The clinically indicated and study-specific scanning time will not exceed 120 minutes.

During the study visits:

* A study team member will review inclusion and exclusion criteria with the participant
* A study team member will review medical history review with the participant
* A safety assessment will occur prior to study procedures
* Study MRI scan
* During which the participant will use an MRI-safe machine to stimulate exercise, similar to pressing a gas pedal

If eligible participants return to CHOP for future clinical imaging, we will also request a study-specific MRI assessment.

ELIGIBILITY:
Inclusion Criteria (Mitochondrial Disease Patients):

* Males and females, between the ages of 7 and 75, inclusive
* Suspected (based on clinical presentation) or definite genetic mitochondrial disease diagnosis (i.e., genetic mutations in the constituents of the mitochondrial respiratory chain and/or genetic mutations that are likely to affect mitochondrial function)
* Clinically eligible for an MRI of the lower leg. We are conducting clinical leg MRI scans of patients with definite mitochondrial disease for indications that include muscle weakness and muscle fatigue.
* Able to perform sub-maximal ankle dorsiflexion leg exercise during the MRI study

Inclusion Criteria (Healthy Controls):

* Males and females, between the ages of 7 and 75 years, inclusive
* Able to perform sub-maximal ankle dorsiflexion leg exercise during the MRI study

Inclusion Criteria (Evaluable Healthy Controls and Cases for Data Analysis):

* To note, we will merge coded datasets from Institutional Review Board (IRB) #15-012445, IRB #16-013364, and IRB #08-006177 with data from this study as part of our data analysis plan.
* Complete and evaluable healthy control and cases from IRB #15-012445, IRB #16-013364, and IRB #08-006177

Exclusion Criteria (Mitochondrial Disease Patients and Healthy Controls):

* In the investigator's opinion, inability to fully comply with research procedures
* Active alcohol and/or substance abuse, including tobacco-use
* A pacemaker; any metal-based medical or non-medical devices/implants; any non-removable metal-based object (e.g., body piercings, jewelry, etc.) that cannot be cleared through radiologic evaluation
* Any history of intraocular injury or fragment in or around the orbit that cannot be cleared through radiologic evaluation
* Any history of bullet, shrapnel, or stabbing wounds that cannot be cleared through radiologic evaluation
* Past or current employment involving (or exposure to) a metal grinder (e.g., at a construction worksite)
* Claustrophobia or any known medical conditions which can be exacerbated by stress, anxiety, or panic attacks triggered by enclosed spaces
* Any potentially interfering clinical MRI contrast agents, as reviewed with the radiology team
* At the discretion of the principal investigator (PI), any medical condition that will interfere with or prevent the safe completion of the study
* Any female participant with childbearing potential who is knowingly pregnant or suspects that she is pregnant will be removed from the study. (Although there are no known risks of MRI on pregnant females or fetuses, there is a possibility of yet undiscovered pregnancy-related risks. Since there is no direct benefit from participating in this protocol for pregnant females, they will be excluded to ensure their long-term safety and that of their unborn fetus.)
* To note, for this protocol, participants are instructed to lie still in the MRI scanner; there is no contrast or sedation. Participants will be asked to perform a brief (< 2 minute) foot-pedal exercise. Investigators will ensure that total MRI scanning time (i.e., clinically indicated and study-specific scanning) does not exceed 120 minutes within a single day. Participants who do not possess the cognitive and/or physical abilities to perform these procedures will not be included.

Exclusion Criteria (Healthy Controls)

* Any history or genetic confirmation of mitochondrial disease

Ages: 7 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of suspected or definite mitochondrial disease patients who are receiving clinical care through the Mitochondrial Medicine Frontier Program
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-exercise CrCEST recovery time (seconds) | During the MRI
  The time it takes after the exercise occurs to recover CrCEST

SECONDARY OUTCOMES:
Resting CrCEST | During the MRI
  Amount of CrCEST prior to exercise
Muscle Lipid Content | During the MRI
  Includes both Intramyocellular lipid (IMCL) and extramyocellular lipids (EMCL) content, both expressed in arbitrary units relative to water signal and relative to creatine
Fat-fraction | During the MRI
  n-point Dixon, expressed as a percentage of the total area

CONTACTS AND LOCATIONS:
Overall Officials: Zarazuela Zolkipli Cunningham, MBChB MRCP, Principal Investigator — Children's Hospital of Phiadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States